CLINICAL TRIAL: NCT02640365
Title: A Phase Ib Dose Escalation Study of MM-398 Plus Irinotecan in Patients With Unresectable Advanced Cancer - DOUBLIRI
Brief Title: A Dose Escalation Study of MM-398 Plus Irinotecan in Patients With Unresectable Advanced Cancer
Acronym: DOUBLIRI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Collaborators: Merrimack Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DOUBLIRI C13-4
Record Dates: First submitted 2015-12-16; First posted 2015-12-28 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Unresectable Advanced Cancer
Keywords: cancer; GERCOR; unresectable; MM-398; CPT-11; colorectal; non colorectal
MeSH Terms: conditions — Neoplasms | interventions — irinotecan sucrosofate; Irinotecan; Leucovorin; Fluorouracil; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GROUP A / GROUP B (two differents cohorts) (Experimental): GROUP A (Patients with unresectable advanced non-colorectal cancer ) - irinotecan + MM-398 dose escalation (3-18 patients)
  Level 1 : initial DOUBLIRI dose 60/90 (0-3 patients)
  * MM-398 : 60mg/m²
  * Irinotecan (CPT-11) : 90mg/m²
  Level 2: DOUBLIRI dose 80/90 (9 - 18 patients)
  * MM-398 : 80mg/m²
  * CPT-11: 90mg/m²
  Level 3A: DOUBLIRI dose 60/120 (12-18 patients)
  * MM-398 : 60mg/m²
  * CPT-11: 120mg/m²
  Level 3B: DOUBLIRI dose : 80/120 (12-18 patients)
  * MM-398 : 80mg/m²
  * CPT-11 : 120 mg/m²
  GROUP B (Patients with unresectable metastatic colorectal cancer)- LV/5FU-bevacizumab+irinotecan+MM-398 dose Escalation (3-18 patients)
  same level as group A + LV/5FU - bevacizumab regimen :
  * Bevacizumab : 5mg/kg(day (d) 1)
  * Leucovorin (LV) : 400mg/m² (d1)
  * 5-fluorouracile infusion (5 FU) :2400mg/m² (d1,2)
  Interventions: Drug: MM-398; Drug: Irinotecan; Drug: Leucovorin (LV); Drug: 5-fluorouracile (5-FU); Drug: bevacizumab

INTERVENTIONS:
Drug: MM-398 — unresectable Advanced non-colorectal cancer
  Other Names: GROUP A
Drug: Irinotecan — unresectable metastatic colorectal cancer
  Other Names: GROUP A
Drug: Leucovorin (LV) — unresectable metastatic colorectal cancer
  Other Names: GROUPE B
Drug: 5-fluorouracile (5-FU) — unresectable metastatic colorectal cancer
  Other Names: GROUPE B
Drug: bevacizumab — unresectable metastatic colorectal cancer
  Other Names: GROUPE B
Drug: MM-398 — unresectable metastatic colorectal cancer
  Other Names: GROUPE B

SUMMARY:
MM-398 (also known as PEP02) is nanoliposomal encapsulated irinotecan: the liposomal formulation is designed to extend plasma circulation and to increase accumulation in the tumor through the enhanced permeability and retention (EPR) effect.

This study introduces a new concept of combining free and nanoliposomal drugs.

DETAILED DESCRIPTION:
This is a dose-finding and therapeutic exploratory phase Ib multi-center, open label study of MM-398 plus irinotecan in two different settings:

* Group A : patients with unresectable advanced non-colorectal cancer who should receive only MM-398 and irinotecan
* Group B : patients with unresectable metastatic colorectal cancer who should receive MM-398 and irinotecan combined with leucovorin, 5-fluorouracil and bevacizumab.

These groups will be enrolling in parallel. Pharmacokinetic and biomarker sampling will also be performed.

There are three periods to this study :

Screening period (up to -28d): patients undergo screening assessments to determine the eligibility for the study

MM-398 treatment period (C1D1 until safety evaluation/progression): patients receive treatment every 2 weeks and undergo biopsies and other required assessments. The treatment period is divided into a maximum of 3 dose levels

Follow up period: patients will be followed-up 30 days after their last dose of MM-398 for final safety assessments, and every 2 months thereafter for overall survival follow-up

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 75 years
2. Histologically proven carcinoma,
3. Documented advanced or metastatic disease not suitable for complete surgical resection
4. Measurable or evaluable lesions according to RECIST v1.1 criteria
5. ECOG performance status 0 - 1
6. Adequate Bone marrow reserves as evidenced by:

   * Absolute Neutrophil Count (ANC) ≥1.5 x 109/L without the use of hematopoietic growth factors
   * platelets ≥ 100 x 109/L
   * hemoglobin > 9 g/dL (may be transfused to maintain or exceed this level)
7. International Normalized Ratio (INR) ≤1.5; aPTT<1.5 x upper normal limit (UNL); EXEMPTION: patients on full anticoagulation therapy due to Venous Thromboembolism (VTE) must have an in-range INR (usually between 2 and 3).
8. Adequate renal function as evidenced by:

   * serum creatinine: < 150µmol/l
   * calculated creatinine clearance > 50ml/min. (recommendation: to be calculated according to the MDRD formula)
9. Total bilirubin < 1.0 x upper normal limit (UNL)
10. Normal ECG or ECG without any clinically significant findings
11. Regular follow-up feasible. A registered patient must be treated and followed at the participating center.
12. Able to understand and sign an informed consent
13. No contraindication to any study drugs
14. Registration in a national health care system (CMU included for France). NB.: prior exposure to irinotecan is allowed, except for irinotecan-refractory patients (i.e. exclusion criteria)

Exclusion Criteria:

1. Active central nervous system metastases (indicated by clinical symptoms, cerebral edema, steroid requirement, or progressive disease)
2. Bone-only disease
3. Clinically significant gastrointestinal (GI) disorder including hepatic disorders, bleeding, inflammation, GI obstruction, or diarrhea > grade 1
4. Patients refractory to irinotecan (i.e. prior exposure to irinotecan-based therapy with progressive disease as best response)
5. Known Dose Limiting Toxicity (DLT) responses to irinotecan
6. Patients known to be homozygous for UGT1A1 *28
7. History of any second malignancy in the last 3 years; patients with prior history of in-situ cancer or basal or squamous cell skin cancer are eligible. Patients with a history of other malignancies are eligible if they have been continuously disease-free for at least 3 years
8. Prior exposure to MM-398
9. Known hypersensitivity to any of the components of MM-398, or other liposomal products
10. Concurrent illnesses that would be a relative contraindication to trial participation such as active cardiac or liver disease

    * Severe arterial thromboembolic events (myocardial infarction, unstable angina pectoris, stroke) less than 6 months before inclusion
    * NYHA Class III or IV congestive heart failure, ventricular arrhythmias
11. Chronic inflammatory bowel disease and/or bowel obstruction
12. Active infection or an unexplained fever >38.5°C during screening visits or on the first scheduled day of dosing (at the discretion of the investigator, patients with tumor fever may be enrolled), which in the investigator's opinion might compromise the patient's participation in the trial or affect the study outcome
13. Prior chemotherapy administered within 3 weeks, or within a time interval less than at least 5 half-lives of the agent, whichever is longer, prior to the first scheduled day of dosing in this study
14. Uncontrolled hypertension (defined as persistent systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg), or history of hypertensive crisis, or hypertensive encephalopathy
15. Received radiation therapy in the last 14 days
16. Major surgery or traumatic injury within the last 28 days
17. Any other medical or social condition deemed by the Investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results including tutelage and guardianship
18. Pregnant or breast feeding; females of child-bearing potential must test negative for pregnancy at the time of enrollment based on a urine or serum pregnancy test. Both male and female patients of reproductive potential must agree to use a reliable method of birth control, during the study and for 6 months following the last dose of study drug.
19. Concomitant administrations use with St John Worth, or CYP3A4 inducing anticonvulsants (phenytoin, Phenobarbital, carbamazepine), ketoconazole, itraconazole, troleandomycin, erythromycin, diltiazem and verapamil
20. Concomitant administration of live attenuated virus vaccine such as yellow fever vaccine
21. Known dihydropyrimidine dehydrogenase (DPD) deficiency
22. Known active hepatitis B or C and/or active or chronic human immunodeficiency virus (HIV)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-11-18 (Actual); Primary Completion 2016-12-07 (Actual); Study Completion 2016-12-07 (Actual)

PRIMARY OUTCOMES:
Adverse Event (AE) | Assessed from study inclusion to 30 days after last dose
Dose Limiting Toxicities (DLT) | DLTs will be evaluated during 28-day period following the first dose of study treatment
Maximal tolerated dose (MTD) | after the last patient in each cohort up to 28 months

SECONDARY OUTCOMES:
Response Rate (RR) | tumor responses will be evaluated every 8 weeks after start treatment up to 29 months
Best overall Response (BOR) | BOR is the best response recorded from the inclusion until treatment failure up to 28 months
Overall survival (OS) | assessed from the date of inclusion to the date of patient death, due to any cause or to the last date the patient was known to be alive, up to 29 months
Progression free survival (PFS) | PFS is the time from the date of inclusion to the date of progressive disease or death up to 29 months
Pharmacokinetic of MM-398 plus irinotecan combination therapy | cycle 1 Day 1 (1 cycle every 2 weeks) at Hour (H) 0, H+1, H+2.5, H+4.5, H+6.5, H+26.5, Day 3, Day 8, Day 15 and 30 days after the last dose of treatment
  to determine the levels of MM-398/irinotecan, SN-38 and SN-38G

CONTACTS AND LOCATIONS:
Overall Officials: Benoist Chibaudel, MD, Study Chair — Franco-British Institute
Locations (1):
- Hôpital Saint Antoine, Paris, France

IPD SHARING:
Plan to Share IPD: No